CLINICAL TRIAL: NCT03707665
Title: Screening Ultrasound Compression Testing in Critically Ill Patients Performed by General Nurses - Validation Study
Brief Title: Deep Venous Thrombosis Screening in the ICU by Nurses
Status: Completed | Type: Observational
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Head physician for science and research, Emergency Medical Service of the Central Bohemian Region, Czech Republic
Other Study IDs: 2018-01
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Deep Venous Thrombosis
Keywords: Compression Ultrasound testing; Nurse
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Compression ultrasound testing — Compression ultrasound testing, screening technique for diagnosing deep venous thrombosis

SUMMARY:
Despite of preventive measures, the incidence of deep venous thrombosis (DVT) in ICU patients is estimated to range from 5-31%. While clinical diagnostics is unreliable, ultrasound compression test (UCT) has proven to be a highly sensitive and specific modality for the recognition of lower extremity DVT. Delegating this competence to ICU nurses can increase UCT availability and enable preventive DVT screening. Therefore, the investigators decided to conduct a clinical study to evaluate the sensitivity and specificity of UCT performed by general ICU nurse in ICU patients compared to an investigation by ICU physician certified in ultrasound. Prior to the study, each nurse-investigator participating in the study undergo one-hour training in UCT and examine 5 patients under supervision. Then, ICU patients without known DVT will be investigated by UCT in the femoral and popliteal region of both lower extremities by trained general ICU nurse-investigators. On the same day, the examination will be repeated by an ICU physician-investigator. The results of the examinations of each patient will be blinded to each other for both investigators until both tests are performed. The sensitivity and specificity of the test performed by general nurse will be calculated in comparison with the examination by a specialist.

ELIGIBILITY:
Inclusion Criteria:

* all ICU patients without known deep venous thrombosis, hospitalised more than 72 hours

Exclusion Criteria:

* contraindication of compression ultrasound testing
* end-of-life decision regimen of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Validity of the compression ultrasound testing in the ICU patients performed by general nurses | One day
  Validity of testing performed by nurses will be compared with investigation by the physician, specialist for compression ultrasound testing

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Department of Anesthesiology, Perioperative Medicine and Intensive Care, J.E. Purkinje University, Masaryk Hospital Usti nad Labem, Usti nad Labem, Czech Republic
Locations (1):
- Emergency Medical Service of the Central Bohemian Region, Beroun, Central Bohemia, Czechia

IPD SHARING:
Plan to Share IPD: No